CLINICAL TRIAL: NCT02480855
Title: Early Identification of People at Risk for Sick-leave Due to Work-related Stress - A Randomized Controlled Study of People With Mental Disorders and Physical Complaints Consulting Primary Health Care
Brief Title: Early Identification of Persons at Risk for Sick-leave Due to Work-related Stress
Acronym: TIDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TIDAS
Record Dates: First submitted 2015-05-20; First posted 2015-06-25 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Occupation-related Stress Disorder
Keywords: work related stress; questionnaire; early identification
MeSH Terms: conditions — Occupational Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Questionnaire and feedback (Other): Patients that will see a doctor randomized to the intervention group will fill in the Work Stress Questionnaire prior to the visit. The doctor gets the results from the questionnaire and then gives consultation to the patient based on the results.
  Interventions: Other: Questionnaire and feedback
- Control group (No Intervention): Patients that will see a doctor randomized to the control group get the usual treatment/consultation and after the visit fill in the Work Stress Questionnaire.

INTERVENTIONS:
Other: Questionnaire and feedback
  Arms: Questionnaire and feedback

SUMMARY:
A vital question for society in general and primary health care in particular is early identification of persons at risk of sickness absence due to work-related stress. Even though both the individual and society can gain a lot from the prevention of absence, not the least since return to work is costly once a person is sick-listed. There is, surprisingly enough, no established method to do this. This project is a randomized controlled study of people with mental disorders and physical complaints consulting primary care. The purpose is to evaluate if a systematic use of early identification of work-related stress, combined with feedback at consultation, at the primary health care centers can prevent sickness absence among employed women and men with common mental disorders and subjective physical health complaints.

DETAILED DESCRIPTION:
There is no method or established practice in primary health care when it comes to the important issue of early identification of people at risk of sickness absence due to work-related stress. But work-related stress is common and can cause ill-health and sick-listing. Therefore it is a vital question for society in general and primary health care in particular finding methods to early identify persons at such risk. Both the individual and society can gain a lot from the prevention of absence, not the least since return to work is costly once a person is sick-listed.

Both women and men see a doctor due to the symptoms, and a majority often goes to the primary health care, and this long before sick-listing comes into question. It could very well be that neither patient, nor doctor is aware that the symptoms the patient describes are caused by work and the stress the patient is subject to there. There is, though, a questionnaire, the Work Stress Questionnaire (WSQ), that has been developed to early identify people at risk.

The purpose of this randomized controlled trial is to evaluate if systematic use of the WSQ can reduce the number of sick-days twelve months on in women and men consulting a primary health care GP due to physical and mental complaints. The intervention consists of giving the GPs the WSQ as a tool for systematic use to early identify people at risk, and then be able to refer the patients to preventive health care and other measures within the primary health care or the patient's occupational health service.

The project will be carried out within the Region Västra Götaland and engage around 40 general practitioners, who will in all recruit 420 participants (210 to intervention group and 210 to control group). A register follow-up on sick-leave, healthcare treatment and the use of medicines will be made 12 months later. Three studies are planned to evaluate the intervention. Yet another study, a focus group study, is planned to make process evaluation of how the participating health care center staff perceive systematic use of the WSQ.

ELIGIBILITY:
Inclusion Criteria:

* Employed women and men, aged 18 - 64 years
* Seeking care for:
* depression
* anxiety
* musculoskeletal disorders
* gastrointestinal and cardio-vascular symptoms
* other stress-related symptoms

Exclusion Criteria:

* Currently on sick-leave or have been on sick-leave with doctor's certificate the last month
* Have been absent from work due to illness more than 7 days the last month (without doctor's certificate)
* On sickness or activity payments
* Pregnant women
* Patients seeking care for:
* allergy
* diabetes
* urinary tract infection
* infections (whooping cough, tonsillitis)
* COPD
* fractures
* lumps and spots
* psychiatric diagnoses such as schizophrenia, other psychoses or bipolar diagnoses
* prolonging of sick-leave certificate
* check up of chronic disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of sick-leave days. | 12 months after inclusion
  Differences in number of sick-leave days between intervention group and control group.
Number of periods of sick-leave, full-time or part-time. | 12 months after inclusion
  Differences in number of sick-leave periods, full-time or part-time between intervention group and control group.

SECONDARY OUTCOMES:
Number of health care treatments. | 12 months after inclusion
  Differences in healthcare treatment between the intervention group and the control group.
Types of health care treatments. | 12 months after inclusion
  Differences in healthcare treatment between the intervention group and the control group.
Number of medicines prescriptions. | 12 months after inclusion
  Differences in the use of medicines between the intervention group and the control group.
Types of medicines prescriptions. | 12 months after inclusion
  Differences in the use of medicines between the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Holmgren, Docent, Principal Investigator — Section for Rehabilitation and Health, Inst for neuro science and physiology, Sahlgrenska academy, University of Gothenburg

REFERENCES:
- [Derived] Hulten AM, Bjerkeli P, Holmgren K. Work-related stress and future sick leave in a working population seeking care at primary health care centres: a prospective longitudinal study using the WSQ. BMC Public Health. 2022 Apr 28;22(1):851. doi: 10.1186/s12889-022-13269-8. PMID 35484592
- [Derived] Hulten AM, Bjerkeli P, Holmgren K. Self-reported sick leave following a brief preventive intervention on work-related stress: a randomised controlled trial in primary health care. BMJ Open. 2021 Mar 22;11(3):e041157. doi: 10.1136/bmjopen-2020-041157. PMID 33753430
- [Derived] Hulten AM, Dahlin-Ivanoff S, Holmgren K. Positioning work related stress - GPs' reasoning about using the WSQ combined with feedback at consultation. BMC Fam Pract. 2020 Sep 11;21(1):187. doi: 10.1186/s12875-020-01258-y. PMID 32917138
- [Derived] Sandheimer C, Hedenrud T, Hensing G, Holmgren K. Effects of a work stress intervention on healthcare use and treatment compared to treatment as usual: a randomised controlled trial in Swedish primary healthcare. BMC Fam Pract. 2020 Jul 6;21(1):133. doi: 10.1186/s12875-020-01210-0. PMID 32631243
- [Derived] Bjerkeli PJ, Skoglund I, Holmgren K. Does early identification of high work related stress affect pharmacological treatment of primary care patients? - analysis of Swedish pharmacy dispensing data in a randomised control study. BMC Fam Pract. 2020 Apr 25;21(1):70. doi: 10.1186/s12875-020-01140-x. PMID 32334516
- [Derived] Holmgren K, Hensing G, Bultmann U, Hadzibajramovic E, Larsson MEH. Does early identification of work-related stress, combined with feedback at GP-consultation, prevent sick leave in the following 12 months? a randomized controlled trial in primary health care. BMC Public Health. 2019 Aug 14;19(1):1110. doi: 10.1186/s12889-019-7452-3. PMID 31412832
- [Derived] Holmgren K, Sandheimer C, Mardby AC, Larsson ME, Bultmann U, Hange D, Hensing G. Early identification in primary health care of people at risk for sick leave due to work-related stress - study protocol of a randomized controlled trial (RCT). BMC Public Health. 2016 Nov 25;16(1):1193. doi: 10.1186/s12889-016-3852-9. PMID 27884137